CLINICAL TRIAL: NCT01183403
Title: Value of Contrast-enhanced Ultrasonography and Magnetic Resonance Enterography to Predict the Efficacy of Anti-TNF Therapy in Crohn's Disease Complicated by Symptomatic Small Bowel Stricture
Brief Title: CE-U and MRE to Predict the Efficacy of Anti-TNF Therapy in Crohn's Disease
Acronym: CREOLE
Status: Completed | Type: Observational
Sponsor: Groupe d'Etude Therapeutique des Affections Inflammatoires Digestives (Other)
Responsible Party: Sponsor
Other Study IDs: GETAID 2008-3
Record Dates: First submitted 2009-09-11; First posted 2010-08-17 (Estimated); Last update posted 2015-06-23 (Estimated); Status verified 2015-06

CONDITIONS: Crohn's Disease
Keywords: stricture; anti-TNF; ileal Crohn'Disease; patients with ileal Crohn's disease complicated by; symptomatic stricture after failure of corticosteroids; and/or immunosuppressives
MeSH Terms: conditions — Crohn Disease; Constriction, Pathologic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The value of anti-TNF therapy in intestinal strictures related to Crohn's disease (CD) has not been clearly demonstrated. The results reported by some teams suggest no beneficial effect or even an increased risk of bowel obstruction in the case of stricture, while other publications indicate a favourable action of anti-TNF in this setting. The efficacy of anti-TNF in patients with intestinal stricture related to Crohn's disease could depend on the lesions responsible for the stricture, as anti-TNF agents are probably effective in inflammatory forms and useless or even potentially harmful in fibrotic forms. In practice, the decision is currently empirical and a trial of anti-TNF therapy is often proposed.

In view of the high incidence of intestinal strictures in CD and the need for a treatment as effective as anti-TNF in this setting, it is important to more clearly define the indications of these treatments guided by the information provided by modern imaging.

The aim of this prospective study is to determine whether certain signs detected by MR enterography and contrast-enhanced ultrasonography can help to predict failure of anti-TNF therapy in patients with CD presenting a symptomatic stricture of the small bowel and scheduled to receive this treatment.

ELIGIBILITY:
Inclusion Criteria:

* Crohn's disease defined according to the usual endoscopic, histological, and radiological criteria
* Small bowel (jejunum or ileum) stricture identified by radiography or endoscopy
* Obstructive symptoms greater than or equal to 3 on a scale from 0 to 6 evaluated over the last 8 weeks
* Failure of corticosteroids and/or immunosuppressives and indication for anti-TNF therapy

Exclusion Criteria:

* Nonresolving complete bowel obstruction
* Previous anti-TNF therapy
* Contraindication to anti-TNF therapy:

  * Intra-abdominal, intra-mural or extramural abscess
  * Active infection
  * Severe infection during the previous 2 months
  * Nontreated latent tuberculosis
  * Heart failure
  * Active malignancy during the previous 5 years
  * Demyelinating neurological disease
* Modification of the treatment of Crohn's disease during the previous two months: azathioprine, mercaptopurine, methotrexate, thalidomide
* Contraindication to MR enterography or contrast-enhanced ultrasonography

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with ileal Crohn's disease complicated by symptomatic stricture after failure of corticosteroids and/or immunosuppressives
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2010-01; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
% of failure defined by the development of at least one of events (obstructive symptoms, activity of the disease..) | 6 months minus baseline

SECONDARY OUTCOMES:
Change of the obstructive symptom scale at the various visits between D0 and W24 | 6 months minus baseline

CONTACTS AND LOCATIONS:
Overall Officials: Yoram BOUHNIK, MD,PhD, Principal Investigator — Groupe d'Etude Therapeutique des Affections Inflammatoires Digestives; Franck CARBONNEL, MD,PhD, Principal Investigator — Groupe d'Etude Therapeutique des Affections Inflammatoires Digestives
Locations (18):
- Ulb - Clinique Saint Luc, Brussels, Belgium
- France (17):
  - Chu Amiens, Amiens
  - Chu Besancon, Besançon
  - Hopital Avicennes, Bobigny
  - Hopital Beaujon, Clichy
  - Hopital Bicetre, Le Kremlin-Bicêtre
  - Chru Lille, Lille
  - Chu Montpellier, Montpellier
  - Chu Nantes, Nantes
  - CHU NICE, Nice
  - Hopital Lariboisiere, Paris
  - Hopital Saint Louis, Paris
  - Hopital St Antoine, Paris
  - Hopital Cochin, Paris
  - Hopital Bichat, Paris
  - Chu Reims, Reims
  - Chu Rouen, Rouen
  - Chu Tours, Tours

REFERENCES:
- [Background] Bernstein CN, Greenberg H, Boult I, Chubey S, Leblanc C, Ryner L. A prospective comparison study of MRI versus small bowel follow-through in recurrent Crohn's disease. Am J Gastroenterol. 2005 Nov;100(11):2493-502. doi: 10.1111/j.1572-0241.2005.00239.x. PMID 16279905
- [Background] Biancone L, Calabrese E, Petruzziello C, Onali S, Caruso A, Palmieri G, Sica GS, Pallone F. Wireless capsule endoscopy and small intestine contrast ultrasonography in recurrence of Crohn's disease. Inflamm Bowel Dis. 2007 Oct;13(10):1256-65. doi: 10.1002/ibd.20199. PMID 17577246
- [Background] Brenner DJ, Hall EJ. Computed tomography--an increasing source of radiation exposure. N Engl J Med. 2007 Nov 29;357(22):2277-84. doi: 10.1056/NEJMra072149. No abstract available. PMID 18046031
- [Background] Chiorean MV, Sandrasegaran K, Saxena R, Maglinte DD, Nakeeb A, Johnson CS. Correlation of CT enteroclysis with surgical pathology in Crohn's disease. Am J Gastroenterol. 2007 Nov;102(11):2541-50. doi: 10.1111/j.1572-0241.2007.01537.x. Epub 2007 Sep 26. PMID 17900329
- [Background] Esteban JM, Aleixandre A, Hurtado MJ, Maldonado L, Mora FJ, Nogues E. Contrast-enhanced power Doppler ultrasound in the diagnosis and follow-up of inflammatory abdominal masses in Crohn's disease. Eur J Gastroenterol Hepatol. 2003 Mar;15(3):253-9. doi: 10.1097/00042737-200303000-00008. PMID 12610320
- [Background] Giorgio A, Ferraioli G, Tarantino L, de Stefano G, Scala V, Scarano F, Coppola C, Del Viscovo L. Contrast-enhanced sonographic appearance of hepatocellular carcinoma in patients with cirrhosis: comparison with contrast-enhanced helical CT appearance. AJR Am J Roentgenol. 2004 Nov;183(5):1319-26. doi: 10.2214/ajr.183.5.1831319. PMID 15505297
- [Background] Guidi L, De Franco A, De Vitis I, Armuzzi A, Semeraro S, Roberto I, Papa A, Bock E, Gasbarrini G, Fedeli G. Contrast-enhanced ultrasonography with SonoVue after infliximab therapy in Crohn's disease. Eur Rev Med Pharmacol Sci. 2006 Jan-Feb;10(1):23-6. PMID 16494107
- [Background] Holtmann M, Wanitschke R, Helisch A, Bartenstein P, Galle PR, Neurath M. [Anti-TNF antibodies in the treatment of inflammatory intestinal stenoses in Crohn's disease]. Z Gastroenterol. 2003 Jan;41(1):11-7. doi: 10.1055/s-2003-36677. German. PMID 12541166
- [Background] Louis E, Boverie J, Dewit O, Baert F, De Vos M, D'Haens G; Belgian IBD Research Group. Treatment of small bowel subocclusive Crohn's disease with infliximab: an open pilot study. Acta Gastroenterol Belg. 2007 Jan-Mar;70(1):15-9. PMID 17619533
- [Background] Masselli G, Brizi GM, Parrella A, Minordi LM, Vecchioli A, Marano P. Crohn disease: magnetic resonance enteroclysis. Abdom Imaging. 2004 May-Jun;29(3):326-34. doi: 10.1007/s00261-003-0116-9. No abstract available. PMID 15354341
- [Background] Masselli G, Casciani E, Polettini E, Gualdi G. Comparison of MR enteroclysis with MR enterography and conventional enteroclysis in patients with Crohn's disease. Eur Radiol. 2008 Mar;18(3):438-47. doi: 10.1007/s00330-007-0763-2. Epub 2007 Sep 25. PMID 17899102
- [Background] Negaard A, Mulahasanovic A, Reisaeter LA, Aasekjaer K, Sandvik L, Klow NE. Crohn's disease evaluated with magnetic resonance enteroclysis: diagnostic performance of experienced and inexperienced readers before and after training. Acta Radiol. 2008 Nov;49(9):967-74. doi: 10.1080/02841850802409539. PMID 18925449
- [Background] Negaard A, Sandvik L, Mulahasanovic A, Berstad AE, Klow NE. Magnetic resonance enteroclysis in the diagnosis of small-intestinal Crohn's disease: diagnostic accuracy and inter- and intra-observer agreement. Acta Radiol. 2006 Dec;47(10):1008-16. doi: 10.1080/02841850600979071. PMID 17135001
- [Background] Parente F, Greco S, Molteni M, Anderloni A, Maconi G, Bianchi Porro G. Modern imaging of Crohn's disease using bowel ultrasound. Inflamm Bowel Dis. 2004 Jul;10(4):452-61. doi: 10.1097/00054725-200407000-00022. PMID 15475759
- [Background] De Pascale A, Garofalo G, Perna M, Priola S, Fava C. Contrast-enhanced ultrasonography in Crohn's disease. Radiol Med. 2006 Jun;111(4):539-50. doi: 10.1007/s11547-006-0049-9. Epub 2006 May 25. English, Italian. PMID 16779540
- [Background] Pelletier AL, Kalisazan B, Wienckiewicz J, Bouarioua N, Soule JC. Infliximab treatment for symptomatic Crohn's disease strictures. Aliment Pharmacol Ther. 2009 Feb 1;29(3):279-85. doi: 10.1111/j.1365-2036.2008.03887.x. Epub 2008 Nov 8. PMID 19035967
- [Background] Di Sabatino A, Fulle I, Ciccocioppo R, Ricevuti L, Tinozzi FP, Tinozzi S, Campani R, Corazza GR. Doppler enhancement after intravenous levovist injection in Crohn's disease. Inflamm Bowel Dis. 2002 Jul;8(4):251-7. doi: 10.1097/00054725-200207000-00003. PMID 12131608
- [Background] Rieder F, Brenmoehl J, Leeb S, Scholmerich J, Rogler G. Wound healing and fibrosis in intestinal disease. Gut. 2007 Jan;56(1):130-9. doi: 10.1136/gut.2006.090456. No abstract available. PMID 17172588
- [Background] Di Sabatino A, Pender SL, Jackson CL, Prothero JD, Gordon JN, Picariello L, Rovedatti L, Docena G, Monteleone G, Rampton DS, Tonelli F, Corazza GR, MacDonald TT. Functional modulation of Crohn's disease myofibroblasts by anti-tumor necrosis factor antibodies. Gastroenterology. 2007 Jul;133(1):137-49. doi: 10.1053/j.gastro.2007.04.069. Epub 2007 May 5. PMID 17631138
- [Background] Sallomi DF. The use of contrast-enhanced power Doppler ultrasound in the diagnosis and follow-up of inflammatory abdominal masses associated with Crohn's disease. Eur J Gastroenterol Hepatol. 2003 Mar;15(3):249-51. doi: 10.1097/00042737-200303000-00007. PMID 12610319
- [Background] Schlottmann K, Kratzer W, Scholmerich J. Doppler ultrasound and intravenous contrast agents in gastrointestinal tract disorders: current role and future implications. Eur J Gastroenterol Hepatol. 2005 Mar;17(3):263-75. doi: 10.1097/00042737-200503000-00003. PMID 15716649
- [Background] Schreyer AG, Geissler A, Albrich H, Scholmerich J, Feuerbach S, Rogler G, Volk M, Herfarth H. Abdominal MRI after enteroclysis or with oral contrast in patients with suspected or proven Crohn's disease. Clin Gastroenterol Hepatol. 2004 Jun;2(6):491-7. doi: 10.1016/s1542-3565(04)00168-5. PMID 15181618
- [Background] Serra C, Menozzi G, Labate AM, Giangregorio F, Gionchetti P, Beltrami M, Robotti D, Fornari F, Cammarota T. Ultrasound assessment of vascularization of the thickened terminal ileum wall in Crohn's disease patients using a low-mechanical index real-time scanning technique with a second generation ultrasound contrast agent. Eur J Radiol. 2007 Apr;62(1):114-21. doi: 10.1016/j.ejrad.2006.11.027. Epub 2007 Jan 18. PMID 17239555
- [Background] Solt J, Hertelendi A, Szilagyi K. [Balloon catheter dilatation of lower gastrointestinal tract stenoses: long-term results]. Orv Hetil. 2002 Aug 4;143(31):1835-40. Hungarian. PMID 12187577
- [Background] Sorrentino D. Role of biologics and other therapies in stricturing Crohn's disease: what have we learnt so far? Digestion. 2008;77(1):38-47. doi: 10.1159/000117306. Epub 2008 Feb 19. PMID 18285676
- [Background] Warnaar N, Hofker HS, Maathuis MH, Niesing J, Bruggink AH, Dijkstra G, Ploeg RJ, Schuurs TA. Matrix metalloproteinases as profibrotic factors in terminal ileum in Crohn's disease. Inflamm Bowel Dis. 2006 Sep;12(9):863-9. doi: 10.1097/01.mib.0000231568.43065.ed. PMID 16954805
- [Derived] Bouhnik Y, Carbonnel F, Laharie D, Stefanescu C, Hebuterne X, Abitbol V, Nachury M, Brixi H, Bourreille A, Picon L, Bourrier A, Allez M, Peyrin-Biroulet L, Moreau J, Savoye G, Fumery M, Nancey S, Roblin X, Altwegg R, Bouguen G, Bommelaer G, Danese S, Louis E, Zappa M, Mary JY; GETAID CREOLE Study Group. Efficacy of adalimumab in patients with Crohn's disease and symptomatic small bowel stricture: a multicentre, prospective, observational cohort (CREOLE) study. Gut. 2018 Jan;67(1):53-60. doi: 10.1136/gutjnl-2016-312581. Epub 2017 Jan 24. PMID 28119352
- See also: Related Info — http://www.getaid.org